CLINICAL TRIAL: NCT05580666
Title: Reducing Mortality in Adults With Advanced HIV Disease, a Double Blinded Randomized Trial
Brief Title: Reducing Mortality in Adults With Advanced HIV Disease (REVIVE)
Acronym: REVIVE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRI.REVIVE
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: HIV Disease Progression
Keywords: Human immunodeficiency virus; Antiretroviral therapy; Azithromycin; Mortality
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Double blinded placebo-controlled randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Azithromycin 250 mg once daily (Experimental): Active Azithromycin tablet
  Interventions: Drug: Azithromycin Oral Tablet
- Oral matching placebo, once daily (Placebo Comparator): Matching placebo tablet
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Azithromycin Oral Tablet — Antimicrobial therapy
  Arms: Oral Azithromycin 250 mg once daily
Drug: Placebo oral tablet — Inert ingredients
  Arms: Oral matching placebo, once daily

SUMMARY:
A double blinded, placebo-controlled, multicenter trial to evaluate effectiveness of azithromycin prophylaxis on mortality in advanced HIV.

DETAILED DESCRIPTION:
All participants in the REVIVE trial will be randomized (1:1) at the time of study entry to receive azithromycin prophylaxis or placebo for 28 days and will be followed for 24 weeks to determine the primary outcome measure. Total follow up duration will be 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Documented HIV infection
3. CD4 count criteria:

   i. CD4 count ≤ 100 cells/mm3 within past 4 weeks; or

   ii. Documented CD4 nadir ≤ 100 cells/mm3 and complete interruption of ART for ≥ 6 months; or

   iii. Documented CD4 count ≤ 100 cells/mm3 if ART-naive
4. Ability to initiate or re-initiate ART, or switch to an effective ART regimen if failing current therapy, within 4 weeks of enrolment

Exclusion Criteria:

1. Contraindications to azithromycin:

   i. Hypersensitivity to azithromycin, erythromycin, or any macrolide antibiotic; or

   ii. Personal or family history of QT-prolongation
2. Severe illness requiring immediate or continued hospitalization (this will be in the judgment of site investigators)
3. Off-label azithromycin prophylaxis or requirement for prolonged (> 7 days) azithromycin (or macrolide) therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 24 weeks after randomization
  All-cause mortality over the first 24 weeks after randomization

SECONDARY OUTCOMES:
All-cause mortality | 12 weeks after randomization
  All-cause mortality over the first 12 weeks after randomization
Hospitalization | 24 weeks after randomization
  Hospitalization over the first 24 weeks after randomization
Composite of hospitalization or all-cause mortality | 24 weeks after randomization
  Composite of hospitalization or all-cause mortality over the first 24 weeks after randomization

CONTACTS AND LOCATIONS:
Overall Officials: John Eikelboom, MBBS, MSc, FRCPC, Principal Investigator — Population Health Research Institute; Sean Wasserman, MBChB, PhD, Principal Investigator — University of Cape Town
Locations (52):
- Côte d’Ivoire (3):
  - Centre Intégré de Recherches Biocliniques d'Abidjan (CIRBA), Abidjan
  - Centre médical de suivi des donneurs de sang (CMSDS), Abidjan
  - Unité de Soins Ambulatoires et de conseils (USAC), Abidjan
- Ethiopia (4):
  - Adama Hospital Medical College, Ādama
  - Asella Referral and Teaching Hospital, Āsela
  - Jimma University Hospital, Jimma
  - Tigray health research institute (THRI), Mek'ele
- Ghana (3):
  - Komfo Anokye Teaching Hospital, Kumasi
  - Kumasi South Hospital, Kumasi
  - Suntreso Government Hospital, Kumasi
- Lilongwe Medical Relief Fund/UNC Project, Lilongwe, Malawi
- Faculty of Medicine, Eduardo Mondlane University, Maputo, Mozambique
- Nigeria (11):
  - University of Abuja Teaching Hospital, Abuja
  - University of Calabar Teaching Hospital, Calabar
  - University of Nigeria Teaching Hospital, Enugu
  - University College Hospital, Ibadan
  - Jos University Teaching Hospital, Jos
  - Aminu Kano Teaching Hospital, Kano
  - Lagos University Teaching Hospital, Lago
  - Usmanu Danfodiyo University Teaching Hos, Sokoto
  - Federal Medical Center, Umuahia
  - University of Uyo Teaching Hospital, Uyo
  - Niger Delta University Teaching Hospital, Yenagoa
- Centre Hospitalier Universitaire de Kigali (CHUK), Kigali, Rwanda
- Sierra Leone (5):
  - 34 Military Hospital, Freetown
  - College of Medicine and Allied Health Sciences, University of Sierra Leone, Freetown
  - Kenema Regional Hospital, Kenema
  - Koidu Government Hospital, Koidu
  - Makeni Regional Hospital, Makeni
- South Africa (16):
  - Desmond Tutu Health Foundation, Cape Town
  - Groote Schuur Hospital -New main building, Infectious Disease Clinic G26, Cape Town
  - New Somerset Hospital, Cape Town
  - Ubuntu Clinic, Site B, Khayelitsha, Wellcome Centre, Cape Town
  - Africa Health Research Institute (AHRI)- Nkundusi Clinic, Hlabisa
  - Africa Health Research Institute (AHRI)- Hluhluwe Clinic, Hluhluwe
  - Wits Health Consortium (Pty) Ltd, Johannesburg
  - The Aurum Institute, Klerksdorp
  - Africa Health Research Institute (AHRI)- KwaMsane Clinic, Mtubatuba
  - Africa Health Research Institute (AHRI)- Mpukunyoni Clinic, Mtubatuba
  - Africa Health Research Institute (AHRI)- Mtubatuba Clinic, Mtubatuba
  - Africa Health Research Institute (AHRI)- Somkhele Clinic, Mtubatuba
  - Livingstone hospital, Port Elizabeth
  - Steve Biko Academic Hospital, University of Pretoria, Pretoria
  - Right to Care NPC, Esizayo Division, Randburg
  - The Aurum Institute, Rustenburg
- Uganda (4):
  - MUJHU, Kampala
  - SICRA Kampala, Kampala
  - SICRA Lira, Lira
  - Mbarara Regional Referral hospital, Mbarara
- Zambia (3):
  - The Center for Infectious Disease Research in Zambia (CIDRZ)- George Clinical Research Site, Lusaka
  - The Center for Infectious Disease Research in Zambia (CIDRZ)- Matero Clinical Research Site, Lusaka
  - The Center for Infectious Disease Research in Zambia (CIDRZ)-Chawama Clinical Research Site (CRS), Lusaka

IPD SHARING:
Plan to Share IPD: No